CLINICAL TRIAL: NCT06749795
Title: A Randomized, Double-Blind, Placebo Controlled, Multi -Center, Phase 1b Study to Evaluate the Safety and Tolerability of LIV001 in Patients with Mild-to-Moderate Active Ulcerative Colitis
Brief Title: LIV001 in Patients with Mild-to-Moderate Active Ulcerative Colitis (UC)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Liveome Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIV001-02
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LIV001 (Experimental): LIV001 will be given orally and daily from baseline until end of study
  Interventions: Drug: LIV001
- Placebo (Placebo Comparator): Placebo will be given orally and daily from baseline until end of study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIV001 — Orally administered for 8 weeks
  Arms: LIV001
Drug: Placebo — Orally administered for 8 weeks
  Arms: Placebo

SUMMARY:
A Phase 1b study to evaluate the safety and tolerability of LIV001 in Patients with Mild-to- Moderate Active Ulcerative Colitis

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, multi-center study to evaluate the safety and tolerability of LIV001 in patients with mild to moderate UC. Patients will receive LIV001 or placebo for 8 weeks. All patients will return to the site for a follow-up visit on week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 years (inclusive) at Screening.
2. Established diagnosis of UC for at least 3 months prior to Screening, diagnosed by routine clinical, radiographic, endoscopic or pathologic criteria (Confirmed by colonoscopy and pathology records or, if unavailable, diagnosis confirmed by a letter from the subject's general practitioner.)

Exclusion Criteria:

1. Possible or confirmed diagnosis of Crohn's Disease, other form of inflammatory bowel disorder and coeliac disease.
2. History of a condition associated with significant immunosuppression, or chronic administration (> 14 consecutive days) of immunosuppressants or other immune-modifying drugs within 3 months prior to Visit 3 (subjects taking oral medications for UC, including corticosteroids or immunomodulators, are not excluded).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2026-01-17 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Baseline through Study Completion (Week 12).
Number of subjects with clinical laboratory abnormalities | Baseline through Study Completion (Week 12).
Number of subjects with changes in the 12-lead electrocardiogram (ECG) | Baseline through Study Completion (Week 12).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Napora, Doctor of Medicine, Principal Investigator — Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska
Locations (1):
- Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No